CLINICAL TRIAL: NCT05261191
Title: A Phase 1 Study of MGD020 as a Single Agent or in Combination With MGD014 in Persons With HIV-1 on Antiretroviral Therapy
Brief Title: A Study of MGD020 Alone or Combined With MGD014 in Persons With HIV-1 on Antiretroviral Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MacroGenics (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institutes of Health (NIH) (NIH); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGD020-01; 272201500032C-P00008-9999-1 (NIH)
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Human Immunodeficiency Virus I Infection; Immunodeficiency Virus Type 1, Human; Human Immunodeficiency Virus Type 1
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1A: Dose level 1 (Experimental): Single dose MGD020
  Interventions: Biological: MGD020
- Part 1A: Dose level 2 (Experimental): Single dose MGD020
  Interventions: Biological: MGD020
- Part 1A: Dose level 3 (Experimental): Single dose MGD020
  Interventions: Biological: MGD020
- Part 1A: Dose level 4 (Experimental): Single dose MGD020
  Interventions: Biological: MGD020
- Part 1A: Dose level 5 (Experimental): Single dose MGD020
  Interventions: Biological: MGD020
- Part 1A: Dose level 6 (Experimental): Single dose MGD020
  Interventions: Biological: MGD020
- Part 1B: MTD/MAD -1 MGD020 and MGD014 (Experimental): Single dose MGD020 and MGD014
  Interventions: Biological: MGD020; Biological: MGD014
- Part 1B: MTD/MAD MGD020 and MGD014 (Experimental): Single dose MGD020 and MGD014
  Interventions: Biological: MGD020; Biological: MGD014
- Part 2: MGD020 and MGD014 (Experimental): Multiple doses of MGD020 and MGD014
  Interventions: Biological: MGD020; Biological: MGD014

INTERVENTIONS:
Biological: MGD020 — MGD020 is a bispecific DART molecule that binds CD3 and gp41 subunit of HIV-1 envelope.
Biological: MGD014 — MGD014 is a bispecific DART molecule that binds CD3 and gp120 subunit of HIV-1 envelope.
  Arms: Part 1B: MTD/MAD -1 MGD020 and MGD014; Part 1B: MTD/MAD MGD020 and MGD014; Part 2: MGD020 and MGD014

SUMMARY:
Study CP-MGD020-01 is a phase 1, open-label, dose-escalation, and multi-dose expansion study of MGD020 as a single agent or in combination with MGD014 in persons with HIV-1 (PWH) on antiretroviral therapy (ART). The study is designed to evaluate the safety, tolerability, pharmacokinetics (PK), immunogenicity, and pharmacodynamics (PD) of the study drugs. The study consists of 3 parts (Part 1A, Part 1B, and Part 2). The participant's standard of care ART regimen is continued throughout the study period.

MGD020 is a bispecific DART® molecule that binds CD3 and gp41 subunit of HIV-1 envelope. MGD014 is a bispecific DART® molecule that binds CD3 and gp120 subunit of HIV-1 envelope. These DART molecules redirect CD3+ T lymphocytes to kill HIV-1-infected CD4+ T cells.

Part 1A evaluates groups of participants given a single dose of MGD020. A 2-week safety period is observed prior to escalation to the next dose level. Dose escalation continues until either the maximum tolerated dose (MTD) or maximum administered dose (MAD) is determined.

Part 1B begins after the end of Part 1A. Part 1B evaluates groups of participants given a single dose of the MGD020 MTD or MAD from Part 1A and a fixed dose of of MGD014. The first group will be treated with a single dose of MGD020, at a dose determined to be one dose lower than the single-agent MTD/MAD from Part 1A, and a single 300 mcg/kg dose of MGD014. Dose escalation proceeds until either the MTD or MAD is determined.

Part 2 begins after the end of Part 1B. Part 2 is a multi-dose expansion group. Each participant will receive the MTD or MAD of MGD020 from Part 1B and a fixed dose of MGD014 from Part 1B, administered every 2 weeks (Q2W) for 3 combination doses over 4 weeks. Up to 6 participants may be enrolled in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years and ≤ 70 years of age and able to provide informed consent
* HIV-1 infection documented by rapid HIV test or HIV enzyme or chemiluminescence immunoassay and confirmed by a different second test.
* Plasma HIV-1 RNA viral load

  * < 50 copies/mL at 2 time points within 24 months prior to screening (1 time point within 12 months prior to screening), and
  * < 50 copies/mL at screening, and
  * Not ≥ 50 copies/mL on 2 consecutive time points within 24 months nor > 1000 copies/mL at any time within 6 months prior to screening
* On continuous antiretroviral therapy (ART) for at least 24 months prior to screening and must continue ART throughout the study.
* CD4 cell count > 350 cells/mm3 at screening
* Acceptable laboratory values related to bone marrow, kidney and liver function.
* Individuals of childbearing potential must agree to use highly effective forms of contraception throughout the study through 6 months after the last dose of MGD014.

Exclusion Criteria:

* History of any HIV-1 vaccine or HIV-1 immunotherapy, except MGD014 or MGD020, within 6 months prior to screening.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient.
* Active viral, bacterial, or systemic fungal infection requiring intravenous antibiotic, antiviral, or antifungal treatment within 7 days prior to the initiation of study drug.
* Active coronavirus disease 19 (COVID-19)/severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection.
* Participation in another investigational clinical research study within 60 days prior to screening.
* History of virologic failure on an ART regimen containing FDA-approved HIV-1 entry inhibitors (maraviroc, enfuvirtide, and/or ibalizumab). Virologic failure is defined as a confirmed plasma HIV-1 RNA ≥ 150 copies/mL following assessment of drug adherence, repeat HIV-1 RNA testing with continued treatment, and/or resistance testing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pepi Pencheva, MD, Study Director — MacroGenics
Locations (3):
- United States (3):
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - UNC Hospital - Chapel Hill, Chapel Hill, North Carolina
  - Case Western Reserve University Hospital, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed treatment in Part 1A or Part 1B may be considered for treatment in a subsequent cohort in Part B2 or Part 2. Participants must continue to meet all eligibility criteria, not have experienced severe adverse events in Part 1, and do not have detectable antidrug antibodies against prior study treatment.
  Subsequent treatments assignments are not defined in advance when entering the study.
Groups:
- Part 1A: Cohort 1: Single dose: 1 mcg/kg MGD020 administered IV
- Part 1A: Cohort 2: Single dose: 3 mcg/kg MGD020 administered IV
- Part 1A: Cohort 3: Single dose: 10 mcg/kg MGD020 administered IV
- Part 1A: Cohort 4: Single dose: 30 mcg/kg MGD020 administered IV
- Part 1A: Cohort 5: Single dose: 100 mcg/kg MGD020 administered IV
- Part 1A: Cohort 6: Single dose: 300 mcg/kg MGD020 administered IV
- Part 1B: Cohort 1: Single dose: 100 mcg/kg MGD020 + 300 mcg/kg MGD014 administered IV.
- Part 1B: Cohort 2: Single dose: 300 mcg/kg MGD020 + 300 mcg/kg MGD014 administered IV.
- Part 2: Three doses: 300 mcg/kg MGD020 + 300 mcg/kg MGD014 administered IV once every 2 weeks for 4 weeks.
Period: Part 1A
Arm/Group | Part 1A: Cohort 1 | Part 1A: Cohort 2 | Part 1A: Cohort 3 | Part 1A: Cohort 4 | Part 1A: Cohort 5 | Part 1A: Cohort 6 | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2
Started | 1 | 1 | 1 | 3 | 3 | 6 | 0 | 0 | 0
Participant Treated in 1A Cohort 2 and Part IB Cohort 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Participant Treated in 1A Cohort 4, 1B Cohort 2 and Part 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Participant Treated in 1A Cohort 4 and Part 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Participant Treated in 1A Cohort 5 and 1B Cohort 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Participant Treated in 1A Cohort 5 and 1B Cohort 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Completed | 1 | 1 | 1 | 3 | 3 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1B
Arm/Group | Part 1A: Cohort 1 | Part 1A: Cohort 2 | Part 1A: Cohort 3 | Part 1A: Cohort 4 | Part 1A: Cohort 5 | Part 1A: Cohort 6 | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0
Participant Treated 1B Cohort 1 and Part 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1A: Cohort 1 | Part 1A: Cohort 2 | Part 1A: Cohort 3 | Part 1A: Cohort 4 | Part 1A: Cohort 5 | Part 1A: Cohort 6 | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1A: Cohort 1 | Part 1A: Cohort 2 | Part 1A: Cohort 3 | Part 1A: Cohort 4 | Part 1A: Cohort 5 | Part 1A: Cohort 6 | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2 | Total
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 6 | 3 | 3 | 3 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline characteristics are reported separately for each cohort.
  years
    Part 1A: number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 6 | 0 | 0 | 0 | 15
    Part 1A | 64.0 (NA) — Standard deviation cannot be calculated for cohort of 1 participant. | 57.0 (NA) — Standard deviation cannot be calculated for cohort of 1 participant. | 50.0 (NA) — Standard deviation cannot be calculated for cohort of 1 participant. | 58.0 (3.46) | 52.0 (14.73) | 53.2 (10.89) |  |  |  | 54.7 (9.39)
    Part 1B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 6
    Part 1B |  |  |  |  |  |  | 59.3 (5.13) | 52.3 (13.32) |  | 55.8 (9.81)
    Part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
    Part 2 |  |  |  |  |  |  |  |  | 57.0 (3.46) | 57.0 (3.46)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline demographics are presented for each cohort in different rows.
  Participants
    Part 1A: number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 6 | 0 | 0 | 0 | 15
    Part 1A: Female | 1 | 0 | 1 | 2 | 1 | 0 |  |  |  | 5
    Part 1A: Male | 0 | 1 | 0 | 1 | 2 | 6 |  |  |  | 10
    Part 1B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 6
    Part 1B: Female |  |  |  |  |  |  | 0 | 1 |  | 1
    Part 1B: Male |  |  |  |  |  |  | 3 | 2 |  | 5
    Part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
    Part 2: Female |  |  |  |  |  |  |  |  | 1 | 1
    Part 2: Male |  |  |  |  |  |  |  |  | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Baseline demographics are reported separately for each cohort.
  Participants
    Part 1A : Asian: number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 6 | 0 | 0 | 0 | 15
    Part 1A : Asian | 0 | 0 | 0 | 0 | 0 | 1 |  |  |  | 1
    Part 1B: Asian: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 6
    Part 1B: Asian |  |  |  |  |  |  | 0 | 0 |  | 0
    Part 2: Asian: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
    Part 2: Asian |  |  |  |  |  |  | 0 |  | 0 | 0
    Part 1A Black or African American: number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 6 | 0 | 0 | 0 | 15
    Part 1A Black or African American | 1 | 0 | 1 | 2 | 2 | 2 |  |  |  | 8
    Part 1B Black or African American: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 6
    Part 1B Black or African American |  |  |  |  |  |  | 1 | 1 |  | 2
    Part 2: Black or African American: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
    Part 2: Black or African American |  |  |  |  |  |  |  |  | 2 | 2
    Part 1A: White: number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 6 | 0 | 0 | 0 | 15
    Part 1A: White | 0 | 1 | 0 | 1 | 1 | 3 |  |  |  | 6
    Part 1B: White: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 6
    Part 1B: White |  |  |  |  |  |  | 1 | 1 |  | 2
    Part 2: White: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
    Part 2: White |  |  |  |  |  |  |  |  | 0 | 0
    Part 1A: American Indian or Alaska Native: number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 6 | 0 | 0 | 0 | 15
    Part 1A: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0
    Part 1B: American Indian or Alaska Native: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 6
    Part 1B: American Indian or Alaska Native |  |  |  |  |  |  | 0 | 1 |  | 1
    Part 2: American Indian or Alaska Native: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
    Part 2: American Indian or Alaska Native |  |  |  |  |  |  |  |  | 0 | 0
    Part 1A: Not Reported: number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 6 | 0 | 0 | 0 | 15
    Part 1A: Not Reported | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0
    Part 1B: Not Reported: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 6
    Part 1B: Not Reported |  |  |  |  |  |  | 1 | 0 |  | 1
    Part 2: Not Reported: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
    Part 2: Not Reported |  |  |  |  |  |  |  |  | 0 | 0
    Part 1A: Other: number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 6 | 0 | 0 | 0 | 15
    Part 1A: Other | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0
    Part 1B: Other: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 6
    Part 1B: Other |  |  |  |  |  |  | 0 | 0 |  | 0
    Part 2: Other: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
    Part 2: Other |  |  |  |  |  |  |  |  | 1 | 1
    Part 1A: Hispanic: number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 6 | 0 | 0 | 0 | 15
    Part 1A: Hispanic | 0 | 0 | 0 | 1 | 0 | 2 |  |  |  | 3
    Part 1B: Hispanic: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 6
    Part 1B: Hispanic |  |  |  |  |  |  | 1 | 2 |  | 3
    Part 2: Hispanic: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
    Part 2: Hispanic |  |  |  |  |  |  |  |  | 2 | 2
    Part 1A: Not Hispanic: number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 6 | 0 | 0 | 0 | 15
    Part 1A: Not Hispanic | 1 | 1 | 1 | 2 | 3 | 4 |  |  |  | 12
    Part 1B: Not Hispanic: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 6
    Part 1B: Not Hispanic |  |  |  |  |  |  | 2 | 1 |  | 3
    Part 2: Not Hispanic: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
    Part 2: Not Hispanic |  |  |  |  |  |  |  |  | 1 | 1
Region of Enrollment [Number; unit: participants] — Population: All participants in Part 1A were enrolled in the United States.
  participants
    United States: number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 6 | 0 | 0 | 0 | 15
    United States | 1 | 1 | 1 | 3 | 3 | 6 |  |  |  | 15
Region of Enrollment [Number; unit: participants] — Population: All participants in Part 1B were enrolled in the United States.
  participants
    United States: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 6
    United States |  |  |  |  |  |  | 3 | 3 |  | 6
Region of Enrollment [Number; unit: participants] — Population: All participants in Part 2 were enrolled in the United States.
  participants
    United States: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
    United States |  |  |  |  |  |  |  |  | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number and Types of Adverse Events (AEs), Including Serious Adverse Events (SAEs), and AEs Leading to Treatment Discontinuation in Participants Receiving MGD020 Alone in Part 1A
Description: Observation of side effects determines the highest safe dose for further study
Time Frame: Throughout the study, up to 43 days
Measure: Number; unit: participants with adverse events by type
Arm/Group | Part 1A: Cohort 1 | Part 1A: Cohort 2 | Part 1A: Cohort 3 | Part 1A: Cohort 4 | Part 1A: Cohort 5 | Part 1A: Cohort 6
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 6
participants with adverse events by type
  Any Adverse Event | 1 | 1 | 1 | 3 | 1 | 5
  Treatment-related Adverse Event | 0 | 1 | 1 | 1 | 0 | 2
  Severe adverse event | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-related severe adverse event | 0 | 0 | 0 | 0 | 0 | 0
  Event leading to MGD020 withdrawal | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number and Types of AEs, Including SAEs, and AEs Leading to Treatment Discontinuation in Participants Receiving MGD020 and MGD014 in Part 1B.
Description: Observation of side effects determines the highest safe dose for further study
Time Frame: Throughout the study, up to 43 days
Measure: Number; unit: participants with AE by type
Arm/Group | Part 1B: Cohort 1 | Part 1B: Cohort 2
Number analyzed (Participants) | 3 | 3
participants with AE by type
  Any AE | 2 | 1
  Treatment-related AE | 2 | 0
  Severe AE | 1 | 0
  Severe treatment-related AE | 0 | 0
  Event leading to MGD020 withdrawal | 0 | 0
  Event leading to MGD014 withdrawal | 0 | 0

3. Primary Outcome: Number and Types of AEs, Including SAEs, and AEs Leading to Treatment Discontinuation in Participants Receiving MGD020 and MGD014 in Part 2.
Description: Observation of side effects determines the highest safe dose for further study
Time Frame: Throughout the study, up to 81 days.
Measure: Number; unit: participants with AE by type
Arm/Group | Part 2
Number analyzed (Participants) | 3
participants with AE by type
  Any AE | 2
  Treatment-related AE | 0
  Severe AE | 0
  Severe treatment-related AE | 0
  Event leading to MGD020 withdrawal | 0
  Event leading to MGD014 withdrawal | 0

4. Secondary Outcome: Mean Maximum Concentration of MGD020
Description: The highest concentration of MGD020 at the end of the infusion
Time Frame: Throughout the study, up to 43 days for Parts 1A and 1B, and up to 78 days for Part 2
Population: All participants who received ay least a single-dose of MGD020, and had at least 1 measurable concentration above the lower limit of quantification (LLOQ). One participant in Part A, cohort 4 was excluded from the analysis due to no measurable concentration above the LLOQ. Mean Cmax for Part 2 is after the third infusion.
Measure: Mean (95% Confidence Interval); unit: mcg/liter
Arm/Group | Part 1A: Cohort 1 | Part 1A: Cohort 2 | Part 1A: Cohort 3 | Part 1A: Cohort 4 | Part 1A: Cohort 5 | Part 1A: Cohort 6 | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 3 | 6 | 3 | 3 | 3
mcg/liter | 54.2 [NA to NA] — Confidence interval cannot be calculated for a cohort = 1. | 45.8 [NA to NA] — Confidence interval cannot be calculated for a cohort = 1. | 185.0 [NA to NA] — Confidence interval cannot be calculated for a cohort = 1. | 540.5 [441.5 to 639.5] | 2000 [1807 to 2193] | 6415 [5729 to 7101] | 3410 [350.5 to 6469] | 6947 [5078 to 8816] | 8593 [7883 to 9303]

5. Secondary Outcome: Mean Maximum Concentration of MGD014
Description: The highest concentration of MGD014 at the end of the infusion (Cmax).
Time Frame: Throughout the study, up to 43 days for Part 1B, and up to 78 days for Part 2
Population: All participants who received at least a single-dose of MGD014, and had at least 1 measurable concentration above the LLOQ. Mean Cmax for Part 2 is after the third infusion.
Measure: Mean (95% Confidence Interval); unit: mcg/liter
Arm/Group | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2
Number analyzed (Participants) | 3 | 3 | 3
mcg/liter | 6070 [4325 to 7815] | 6297 [5213 to 7380] | 7043 [6694 to 7393]

6. Secondary Outcome: Mean Time to Maximal Concentration of MGD020
Description: The amount of time required to get maximum concentration of MGD020
Time Frame: Throughout the study, up to 43 days for Parts 1A and 1B, and up to 78 days for Part 2
Population: All participants who received at least a single-dose of MGD020, and had at least 1 measurable concentration above the LLOQ. One participant in Part A, cohort 4 was excluded from the analysis due to no measurable concentration above the LLOQ.. Mean Tmax for Part 2 is after the first infusion.
Measure: Mean (Full Range); unit: hours
Arm/Group | Part 1A: Cohort 1 | Part 1A: Cohort 2 | Part 1A: Cohort 3 | Part 1A: Cohort 4 | Part 1A: Cohort 5 | Part 1A: Cohort 6 | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 3 | 6 | 3 | 3 | 3
hours | 1.4 [NA to NA] — Full range is not applicable to a cohort of 1. | 2.1 [NA to NA] — Full range is not applicable to a cohort of 1. | 2.1 [NA to NA] — Full range is not applicable to a cohort of 1. | 1.6 [1.1 to 2.0] | 1.4 [1.1 to 2.0] | 2.1 [1.1 to 5.0] | 3.8 [1.1 to 6.6] | 1.2 [1.0 to 1.4] | 1.0 [1.0 to 1.0]

7. Secondary Outcome: Mean Time to Maximal Concentration of MGD014
Description: The amount of time required to get maximum concentration of MGD014
Time Frame: Throughout the study, up to 43 days for Part 1B, and up to 78 days for Part 2
Population: All participants who received at least a single-dose of MGD014, and had at least 1 measurable concentration above the LLOQ. Mean Tmax for Part 2 is after the first infusion.
Measure: Mean (Full Range); unit: hours
Arm/Group | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2
Number analyzed (Participants) | 3 | 3 | 3
hours | 2.7 [1.1 to 5.1] | 1.7 [1.0 to 2.1] | 1.3 [1.0 to 2.0]

8. Secondary Outcome: Mean Area Under the Concentration-time Curve (AUC) of MGD020
Description: Total body exposure to MGD020
Time Frame: Throughout the study, up to 43 days for Parts 1A and 1B, and up to 78 days for Part 2
Population: All participants who received at least a single-dose of MGD020, and had at least 1 measurable concentration above the LLOQ. One participant in Part A, cohort 4 was excluded from the analysis due to no measurable concentration above the LLOQ. Mean AUC for Part 2 is after the first infusion.
Measure: Mean (95% Confidence Interval); unit: mcg*hour/liter
Arm/Group | Part 1A: Cohort 1 | Part 1A: Cohort 2 | Part 1A: Cohort 3 | Part 1A: Cohort 4 | Part 1A: Cohort 5 | Part 1A: Cohort 6 | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 3 | 6 | 3 | 3 | 3
mcg*hour/liter | 5570 [NA to NA] — CI cannot be calculated for cohort = 1. | 9280 [NA to NA] — CI cannot be calculated for cohort = 1. | 29400 [NA to NA] — CI cannot be calculated for cohort = 1. | 88900 [63224 to 114576] | 283667 [213313 to 354021] | 957833 [804523 to 1111143] | 365667 [311299 to 420035] | 1088333 [790851 to 1385815] | 854333 [771129 to 937538]

9. Secondary Outcome: Mean AUC of MGD014
Description: Total body exposure to MGD014
Time Frame: Throughout the study, up to 43 days for Parts 1B, and up to 78 days for Part 2
Population: All participants who received at least a single-dose of MGD014, and had at least 1 measurable concentration above the LLOQ. Mean AUC for Part 2 is after the first infusion.
Measure: Mean (95% Confidence Interval); unit: mcg*hour/liter
Arm/Group | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2
Number analyzed (Participants) | 3 | 3 | 3
mcg*hour/liter | 572333 [516478 to 628189] | 631000 [458086 to 803914] | 581333 [511390 to 651276]

10. Secondary Outcome: Mean Half-life of MGD020
Description: The amount of time needed for the body to clear half of the dose of MGD020
Time Frame: Throughout the study, up to 43 days for Parts 1A and 1B, and up to 78 days for Part 2
Population: All participants who received at least a single-dose of MGD020, and had at least 1 measurable concentration above the LLOQ. One participant in Part A, cohort 4 was excluded from the analysis due to no measurable concentration above the LLOQ.. Mean half-life for Part 2 is after the third infusion.
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Part 1A: Cohort 1 | Part 1A: Cohort 2 | Part 1A: Cohort 3 | Part 1A: Cohort 4 | Part 1A: Cohort 5 | Part 1A: Cohort 6 | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 3 | 6 | 3 | 3 | 3
hours | 202 [NA to NA] — CI cannot be calculated for a cohort of 1. | 462 [NA to NA] — CI cannot be calculated for a cohort of 1. | 209 [NA to NA] — CI cannot be calculated for a cohort of 1. | 309 [219 to 398] | 323 [229 to 418] | 221 [94.0 to 348] | 353 [238 to 468] | 361 [322 to 401] | 452 [430 to 475]

11. Secondary Outcome: Mean Half-life of MGD014
Description: The amount of time needed for the body to clear half of the dose of MGD014
Time Frame: Throughout the study, up to 43 days for Parts 1B, and up to 78 days for Part 2
Population: All participants who received at least a single-dose of MGD014, and had at least 1 measurable concentration above the LLOQ. Mean AUC for Part 2 is after the third infusion.
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2
Number analyzed (Participants) | 3 | 3 | 3
hours | 273 [179 to 368] | 296 [287 to 314] | 339 [325 to 353]

12. Secondary Outcome: Mean Volume of Distribution at Steady State (Vss) of MGD020
Description: This parameter measures how much of the drug remains in the bloodstream or is distributed to body tissues.
Time Frame: Throughout the study, up to 78 days for Part 2
Population: Only participants who received at least 3 doses of MGD020 can be evaluated for Vss. All other cohorts receive only 1 dose, so Vss cannot be calculated in Parts 1A and 1B. Vss is reported only for Part 2 after the third dose of MGD020.
Measure: Mean (95% Confidence Interval); unit: liters
Groups:
- Part 1A: Cohort 3: Single dose: 3 10 mcg/kg MGD020 administered IV
Arm/Group | Part 1A: Cohort 1 | Part 1A: Cohort 2 | Part 1A: Cohort 3 | Part 1A: Cohort 4 | Part 1A: Cohort 5 | Part 1A: Cohort 6 | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
liters |  |  |  |  |  |  |  |  | 4.0 [3.5 to 4.6]

13. Secondary Outcome: Mean Volume of Distribution at Steady State of MGD014
Description: This parameter measures how much of the drug remains in the bloodstream or is distributed to body tissues.
Time Frame: Throughout the study, up to 78 days for Part 2
Population: Only participants who received at least 3 doses of MGD014 can be evaluated for Vss. All other cohorts receive only 1 dose, so Vss cannot be calculated in Parts 1A and 1B. Vss is reported only in Part 2 after the third dose of MGD014.
Measure: Mean (95% Confidence Interval); unit: liters
Arm/Group | Part 1A: Cohort 1 | Part 1A: Cohort 2 | Part 1A: Cohort 3 | Part 1A: Cohort 4 | Part 1A: Cohort 5 | Part 1A: Cohort 6 | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
liters |  |  |  |  |  |  |  |  | 3.5 [2.8 to 4.2]

14. Secondary Outcome: Mean Clearance of MGD020
Description: Total body clearance of the drug from plasma of MGD020
Time Frame: Throughout the study, up to 43 days for Parts 1A and 1B, and up to 78 days for Part 2
Population: All participants who received at least a single-dose of MGD020, and had at least 1 measurable concentration above the LLOQ. One participant in Part A, cohort 4 was excluded from analysis due to no measurable concentration above the LLOQ.
Measure: Mean (95% Confidence Interval); unit: liters
Arm/Group | Part 1A: Cohort 1 | Part 1A: Cohort 2 | Part 1A: Cohort 3 | Part 1A: Cohort 4 | Part 1A: Cohort 5 | Part 1A: Cohort 6 | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 3 | 6 | 3 | 3 | 3
liters | 0.02 [NA to NA] — CI cannot be calculated for a cohort of 1. | 0.03 [NA to NA] — CI cannot be calculated for a cohort of 1. | 0.04 [NA to NA] — CI cannot be calculated for a cohort of 1. | 0.03 [0.02 to 0.04] | 0.034 [0.034 to 0.035] | 0.03 [0.02 to 0.03] | 0.03 [0.02 to 0.03] | 0.02 [0.01 to 0.03] | 0.012 [0.011 to 0.013]

15. Secondary Outcome: Mean Clearance of MGD014
Description: Total body clearance of the drug from plasma of MGD014
Time Frame: Throughout the study, up to 43 days for Parts 1B, and up to 78 days for Part 2
Population: All participants who received at least one dose of MGD014. Clearance for Part 2 is reported after the third dose of MGD014.
Measure: Mean (95% Confidence Interval); unit: liters
Arm/Group | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2
Number analyzed (Participants) | 3 | 3 | 3
liters | 0.02 [0.01 to 0.02] | 0.04 [0.02 to 0.05] | 0.02 [0.015 to 0.02]

16. Secondary Outcome: Number of Participants With Elevations in Serum Cytokine Levels of IFN-γ, IL-2, IL-5, IL-6, IL-10, or TNF-α
Time Frame: Throughout the study, up to 43 days for Parts 1A and 1B, and up to 78 days for Part 2.
Population: All participants who received at least one dose of assigned study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: Cohort 1 | Part 1A: Cohort 2 | Part 1A: Cohort 3 | Part 1A: Cohort 4 | Part 1A: Cohort 5 | Part 1A: Cohort 6 | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 6 | 3 | 3 | 3
Participants
  No elevation of serum cytokine levels | 1 | 1 | 1 | 3 | 3 | 3 | 1 | 1 | 0
  Elevation of at least 1 serum cytokine level. | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 3

17. Secondary Outcome: Anti-drug Antibody Formation to MGD020
Description: Number of patients who develop antibodies against MDG020
Time Frame: Throughout the study, up to 43 days for Parts 1A and 1B, and up to 78 days for Part 2
Population: All participants who received at least one dose of assigned study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: Cohort 1 | Part 1A: Cohort 2 | Part 1A: Cohort 3 | Part 1A: Cohort 4 | Part 1A: Cohort 5 | Part 1A: Cohort 6 | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 6 | 3 | 3 | 3
Participants
  Negative before treatment and negative after treatment | 1 | 0 | 1 | 3 | 3 | 4 | 3 | 3 | 3
  Negative before treatment and positive at least once after treatment | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Positive before treatment and positive after treatment | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0

18. Secondary Outcome: Anti-drug Antibody Formation to MGD014
Description: Number of patients who develop antibodies against MDG014
Time Frame: Throughout the study, up to 43 days for Parts 1B, and up to 78 days for Part 2
Population: All participants who received at least 1 dose of MGD014. Participants in Part 1A did not receive MGD014.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2
Number analyzed (Participants) | 3 | 3 | 3
Participants
  Negative before treatment, and negative after treatment | 3 | 3 | 3
  Negative before treatment, and positive at least once after treatment | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The safety assessment is based on evaluation of AEs occurring from the first administration of study drug(s) through the End of Study Visit or 30 days after the last dose of study drug(s) [up to approximately Day 43 in Part 1A and 1B, and up to approximately 81 days in Part 2] , whichever is later. The safety assessment is based on signs, symptoms, physical examination findings, and laboratory test results.
Groups:
- Part 1A: Cohort 1: Single dose: 1 mcg/kg MGD-020 administered IV
- Part 1A: Cohort 2: Single dose: 3 mcg/kg MGD-020 administered IV
- Part 1A: Cohort 3: Single dose: 10 mcg/kg MGD-020 administered IV
- Part 1A: Cohort 4: Single dose: 30 mcg/kg MGD-020 administered IV
- Part 1A: Cohort 6: Single dose: 300 mcg/kg MGD-020 administered IV
- Part 1B: Cohort 1: Single dose: 100 mcg/kg MGD-020 + 300 mcg/kg MGD014 administered IV.
- Part 1B: Cohort 2: Single dose: 300 mcg/kg MGD-020 + 300 mcg/kg MGD014 administered IV.
- Part 2: Three doses: 300 mcg/kg MGD-020 + 300 mcg/kg MGD014 administered IV once every 2 weeks for 4 weeks.
Arm/Group | Part 1A: Cohort 1 | Part 1A: Cohort 2 | Part 1A: Cohort 3 | Part 1A: Cohort 4 | Part 1A: Cohort 5 | Part 1A: Cohort 6 | Part 1B: Cohort 1 | Part 1B: Cohort 2 | Part 2
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/3 | 0/3 | 0/6 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/3 | 0/3 | 0/6 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 3/3 | 1/3 | 5/6 | 2/3 | 1/3 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A: Cohort 1 (N=1) | Part 1A: Cohort 2 (N=1) | Part 1A: Cohort 3 (N=1) | Part 1A: Cohort 4 (N=3) | Part 1A: Cohort 5 (N=3) | Part 1A: Cohort 6 (N=6) | Part 1B: Cohort 1 (N=3) | Part 1B: Cohort 2 (N=3) | Part 2 (N=3)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Visual field defect (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pustule (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vascular access site vesicles (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Carbon dioxide decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0
Brain fog (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT05261191/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT05261191/SAP_001.pdf